CLINICAL TRIAL: NCT04676815
Title: Application of Narrow Band Imaging (NBI) Under Electronic Bronchoscope in the Diagnosis and Staging of Lung Cancer
Brief Title: Narrow Band Imaging (NBI) Under Electronic Bronchoscope in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Associate Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: YHe
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Malignant Airway Obstruction
MeSH Terms: conditions — Lung Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NBI PATIENT: Diagnostic Test: NBI in combination with electronic bronchoscope
  Interventions: Procedure: NBI and interventional bronchoscopy
- Non-NBI PATIENT: Diagnostic Test: Electronic bronchoscope without NBI

INTERVENTIONS:
Procedure: NBI and interventional bronchoscopy — NBI used to enhance the contrast between the mucosal surface and underlying blood vessels
  Groups: NBI PATIENT

SUMMARY:
Narrow-Band Imaging (NBI) is useful to better demarcate the superficial extent of central type of lung cancer, but its sensitivity and specificity in clinical practice were little studied. This study aimed to investigate the diagnostic effects of NBI in suspected patients with central lung cancer and its application in staging diagnosis of central lung cancer.

DETAILED DESCRIPTION:
With high morbidity and mortality, lung cancer is one of the most common tumors in the world. Therefore, early detection, accurate diagnosis and staging division can effectively guide clinical interventions, thereby improving patient survival. Narrowband imaging under electronic bronchoscope (NBI) is an emerging optical image emphasis technology that can enhance the contrast between the mucosal surface and underlying blood vessels, specifically display the distribution of blood vessels, and highlight the subtle changes in mucosal structure. Meanwhile, it can reduce unnecessary biopsy with low risk and costs. In recent years, NBI technology has gradually begun to show its unique advantages in the diagnosis of gastric cancer, esophageal cancer, nasopharyngeal cancer, and bladder cancer. The purpose of this study is to explore the diagnostic value of NBI under electronic bronchoscopy for early detection and accurate diagnosis of lung cancer, and to provide a more economical, safer and more efficient diagnosis option for lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients had a history or current central lung cancer

Exclusion Criteria:

- NONE

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIGH RISK OF CENTRAL TYPE OF LUNG CANCER
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The specificity of diagnosis of NBI plus electronic bronchoscopy in central type lung cancer | 4 months
  Abnormal blood vessels or lack of staining is defined as suspected lesions. All the suspected lesions were biopsied.

SECONDARY OUTCOMES:
The sensitivity, positive predictive value, and negative predictive value. | 4 months
  Abnormal blood vessels or lack of staining is defined as suspected lesions. All the suspected lesions were biopsied.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wen S, Dai L, Wang L, Wang W, Wu D, Wang K, He Z, Wang A, Chen H, Zhang P, Dong X, Dong YA, Wang K, Yao M, Wang M. Genomic Signature of Driver Genes Identified by Target Next-Generation Sequencing in Chinese Non-Small Cell Lung Cancer. Oncologist. 2019 Nov;24(11):e1070-e1081. doi: 10.1634/theoncologist.2018-0572. Epub 2019 Mar 22. PMID 30902917
- [Result] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Result] Subramanian V, Ragunath K. Advanced endoscopic imaging: a review of commercially available technologies. Clin Gastroenterol Hepatol. 2014 Mar;12(3):368-76.e1. doi: 10.1016/j.cgh.2013.06.015. Epub 2013 Jun 28. PMID 23811245
- [Result] Ueda T, Dohi O, Naito Y, Yoshida T, Azuma Y, Ishida T, Matsumura S, Kitae H, Takayama S, Mizuno N, Nakano T, Iwai N, Hirose R, Inoue K, Yoshida N, Kamada K, Uchiyama K, Ishikawa T, Takagi T, Konishi H, Nishimura A, Kishimoto M, Itoh Y. Diagnostic performance of magnifying blue laser imaging versus magnifying narrow-band imaging for identifying the depth of invasion of superficial esophageal squamous cell carcinoma. Dis Esophagus. 2021 Mar 8;34(3):doaa078. doi: 10.1093/dote/doaa078. PMID 32691042
- [Result] Ueyama H, Kato Y, Akazawa Y, Yatagai N, Komori H, Takeda T, Matsumoto K, Ueda K, Matsumoto K, Hojo M, Yao T, Nagahara A, Tada T. Application of artificial intelligence using a convolutional neural network for diagnosis of early gastric cancer based on magnifying endoscopy with narrow-band imaging. J Gastroenterol Hepatol. 2021 Feb;36(2):482-489. doi: 10.1111/jgh.15190. Epub 2020 Jul 28. PMID 32681536